CLINICAL TRIAL: NCT04467580
Title: Development and Validation of an Inflammation Index (FILM-i) and a Fibrosis Index (FILM-f), Combining MRI and Positron Emission Tomography (PET) With Low-dose [18F]FDG (With the Tracer Fluorine-18 (18F) Fluorodeoxyglucose (FDG), Called [18F]FDG PET Activity, to Characterize Fibrosis and Inflammation of Intestinal Strictures During Crohn's Disease
Brief Title: Development of Inflammation and Fibrosis Index, Combining MRI and PET 18F-FDG, in Patient's With Crohn's Disease
Acronym: FILM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020_003067-26
Record Dates: First submitted 2020-06-22; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patient with stenosing CD and for which the surgical resection of one or more stenosis (s) of the terminal ileum is programmed as part of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with stenosing CD (Experimental): Patients with stenosing CD will be recruited in each investigation center, during a preoperative consultation for an already decided and planned intestinal resection (digestive surgery or hepato-gastro department) -enterology).
  Interventions: Diagnostic Test: abdominal [18F]FDG PET/CT

INTERVENTIONS:
Diagnostic Test: abdominal [18F]FDG PET/CT — Patients will have within a maximum period of 15 days before the surgery (resection of intestinal stenosis), records by MRI and by digital PET/CT with low injected activity of [18F]FDG, focused on the abdomen, the MRI will be performed maximum 30 days before the intervention (if available and performed according to the procedure for the study, it will not be repeated for the study).

SUMMARY:
Chronic inflammatory bowel disease (IBD) is a disabling, incurable condition that affects 250,000 people in France, and Crohn's disease (CD) is the most common form. CD progresses, in one-quarter of the cases, towards the appearance of intestinal stenosis, most often on the terminal ileum, sometimes with obstructive symptoms and requiring an optimization of medical treatment (biotherapies) and/or surgery The hypothesis of this study is [18F]FDG PET /CT, (Positron emission tomography with the tracer fluorine-18 (18F) fluorodeoxyglucose (FDG), called [18F]FDG PET coupled to a dedicated CT scanner) could help quantify intestinal inflammation in patients with abnormal entero-MRI, and differentiate inflammation and fibrosis on a joint PET /CT and MRI , in patients with complicated Crohn Disease intestinal stenosis

DETAILED DESCRIPTION:
Intestinal inflammation could be quantified by the PET/CT due to the tropism of a PET tracer, [18F]FDG for activated inflammatory cells.

[18F]FDG PET/CTperformed on latest digital PET/CT cameras and recordings focused on the abdomen could help quantify intestinal inflammation in patients with abnormal entero-MRI, and differentiate inflammation and fibrosis on a joint PET/CT and MRI , in patients with complicated Crohn Disease intestinal stenosis.

Magnetic resonance imaging (MRI) indices are used to assess the upgradability and activity of CD and try to predict response to treatment, in particular Nancy's MRI score for digestive inflammation.

An inflammation index (FILM-i) and a fibrosis index (FILM-f), based on this MRI/PET analysis, will be developed and validated to develop personalized medicine in patients with stenosing CD. Indeed, these indices will guide the therapeutic choice, in particular for the biotherapies prescription or the need to operate these patients.

ELIGIBILITY:
Inclusion Criteria:

* Major subject having received complete information of the clinical research and having signed their informed consent
* Subject with a stenosing CD (objectified on MRI, CT and / or endoscopy).
* Subject for which surgical resection of one or more stenosis (s) of the terminal ileum is programmed as part of the treatment.
* Subject with a social security scheme

Exclusion Criteria:

* Subject having a contraindication to performing MRI and / or PET / CT at 18F-FDG.
* Subject with an ostomy
* Diabetic subject treated by metformin.
* Subject referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code.
* Pregnant woman, parturient or nursing mother.
* Subject with a legal protection measure (guardianship, curatorship, safeguard of justice).
* Subject unable to express consent.
* Subject deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under articles L. 3212-1 and L.3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-05-02 (Estimated)

PRIMARY OUTCOMES:
Index FILM-i | Day 45
  Index FILM-i will be developed using histological scores determined according to the extent and the diffusion in the thickness of the intestinal wall: cellular infiltration and edema
  These histological scores both include 4 grades:
  * 0 = no damage (fibrosis or inflammation),
  * 1 = slight damage,
  * 2 = average achievement,
  * 3 = severe damage. The FILM-i indice is developed in order to predict these same 4 grades.
Index FILM-f | Day 45
  Index FILM-f will be developed using histological scores determined according to the extent and the diffusion in the thickness of the intestinal wall : collagen fibrosis
  These histological scores both include 4 grades:
  * 0 = no damage (fibrosis or inflammation),
  * 1 = slight damage,
  * 2 = average achievement,
  * 3 = severe damage. The FILM-i indice is developed in order to predict these same 4 grades.

SECONDARY OUTCOMES:
Contribution of [18F]FDG PET/CT with index NET (Net Reclassification Index) | Day 45
  Quantify the contribution of [18F]FDG PET/CT, in addition to MRI, for the characterization of the fibrotic and inflammatory components of stenosis of the terminal ileum with the index NET. This index will be calculated to quantify the contribution of PET items to the model including only MRI items.
To compare the performance of the inflammation index (FILM-i) with that of a baseline MRI score, the Nancy score, for the detection of significant colonic inflammation (moderate to severe in histopathology). | Day 45
  The performance of the FILM-i index and Nancy's score will be evaluated by the of correctly classified segments.
Inter- and intra-observer reproducibility | Day 45
  To estimate the inter- and intra-observer reproducibility of the 4 grade classifications obtained by the FILM-i and FILM-f indices with the intra-class correlation coefficients.
Degree of correlation between FILM-i and FILM-f index and the modified histological activity score of the Global Histologic Activity Score (GHAS). | Day 45
  Compare the results of index and modified GHAS score